CLINICAL TRIAL: NCT02764970
Title: Heart Rate Reducing Therapy With Ivabradine and Bisoprolol Before Coronary Computer Tomographic Angiography in Ambulant Patients
Brief Title: Heart Rate Reducing Therapy in Cardiac CT Using Ivabradine and Bisoprolol
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 26-130 ex 13/14
Record Dates: First submitted 2016-03-15; First posted 2016-05-06 (Estimated); Results first posted 2018-03-19 (Actual); Last update posted 2018-03-19 (Actual); Status verified 2017-08

CONDITIONS: Bradycardia
MeSH Terms: conditions — Bradycardia | interventions — Ivabradine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ivabradine 7.5mg orally: patients are pretreated with ivabradine and bisoprolol orally before Cardiac CT angiogram
  Interventions: Drug: Ivabradine 7.5mg orally
- bisoprolol: patients are only pretreated with bisoprolol orally before Cardiac CT angiogram

INTERVENTIONS:
Drug: Ivabradine 7.5mg orally — additive use to the standard medication with bisoprolol
  Other Names: ivabradine is marketed as Procoralan
  Groups: ivabradine 7.5mg orally

SUMMARY:
Out-patients scheduled for coronary computer tomographic angiography (CCTA) were screened regarding their baseline heart rate. If heart rate was > 75, patients were pretreated with 10mg bisoprolol (group 1) or 10mg bisoprolol plus 7.5mg ivabradine (group 2) to reduce heart rate one our before CCTA was performed.

Heart rate, additional use of i.v. bradycardic agents, motion artefacts, radiation dose and drug tolerance was monitored.

DETAILED DESCRIPTION:
Aim of the study is to evaluate if ivabradine, an inhibitor of the funny channel (If), in addition to bisoprolol is effective in lowering heart rate before coronary computer tomographic angiography (CCTA) if administered orally one hour before the scan.

Out-patients of a single radiology center are included in this retrospective analysis. All patients are referred to an ambulant CCTA. All scans are performed with a Siemens Somatom Sensation Cardiac 64 Computer Tomograph and analyzed with Siemens Syngo Plaza software. Patients with an initial heart rate of ≥ 75 bpm are either pretreated with bisoprolol 10mg p.o. alone (group 1) or a combination of bisoprolol 10mg and ivabradine 7.5mg p.o. (group 2) one hour before the CT scan.

The change in treatment from bisoprolol only to the combination of bisoprolol and ivabradine was introduced as a change in standard treatment independent of the study. The study was only plannend and performed as a retrospective analysis after the last patient included into the analysis was already treated.

Additional betablocker is administered intravenously right before the scan if heart rate remains elevated.

The hypothesis is that the addition of ivabradine to bisoprolol results in a pronounced heart rate reduction. This heart rate reduction will lead to a reduced need of i.v. bradicardic drug use, a reduction in motion artifacts and a reduced radiation dose to to a higher rate of flash sequences.

ELIGIBILITY:
Inclusion Criteria:

* all comer study

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients presenting at the radiology center for a planned coronary computer tomographic angiography
Sampling Method: Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2015-02; Primary Completion 2015-09 (Actual); Study Completion 2016-01 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ivabradine 7.5mg Orally | Bisoprolol
Started | 65 | 47
Completed | 65 | 47
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ivabradine 7.5mg Orally | Bisoprolol | Total
Number analyzed (Participants) | 65 | 47 | 112
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 40 | 22 | 62
  >=65 years | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (11) | 63 (10) | 61 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 23 | 49
  Male | 39 | 24 | 63
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Austria | 65 | 47 | 112
heart rate [Mean (Standard Deviation); unit: beats per minute] | 84.1 (6.7) | 80.7 (5.1) | 82.8 (5.0)

OUTCOME MEASURES:

1. Primary Outcome: Heart Rate
Description: number of beats per minute
Time Frame: intraoperative
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Ivabradine 7.5mg Orally | Bisoprolol
Number analyzed (Participants) | 65 | 47
beats per minute | 65.1 (9.8) | 62.7 (9.1)

2. Secondary Outcome: Number of Participants With Use of i.v. Betablocker
Description: measured in mg metoprolol used
Time Frame: time from first ECG in the CT-room to start of CT scan (average of 10 minutes)
Measure: Number; unit: participants
Arm/Group | Ivabradine 7.5mg Orally | Bisoprolol
Number analyzed (Participants) | 65 | 47
participants | 19 | 17

3. Secondary Outcome: Radiation Dose
Description: as calculated in mSv
Time Frame: intraoperative
Measure: Mean (Standard Deviation); unit: mSv
Arm/Group | Ivabradine 7.5mg Orally | Bisoprolol
Number analyzed (Participants) | 65 | 47
mSv | 12.9 (3.4) | 13.2 (3.6)

4. Secondary Outcome: Motion Artifacts
Description: Counted linear misalignments in the ap projection
Time Frame: intraoperative
Measure: Mean (Standard Deviation); unit: linear misalignments in the ap projectio
Arm/Group | Ivabradine 7.5mg Orally | Bisoprolol
Number analyzed (Participants) | 65 | 47
linear misalignments in the ap projectio | 5 (3.2) | 3.5 (4.4)

ADVERSE EVENTS:
Time Frame: 2 hours
Description: Clinically significant bradycardia, hypotension and dizziness were checked
Arm/Group | Ivabradine 7.5mg Orally | Bisoprolol
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/47
Other Adverse Events (participants affected / at risk) | 0/65 | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes